CLINICAL TRIAL: NCT01354132
Title: Effects of Oral N-Acetyl-Cysteine (NAC) in the Early Phase of Schizophrenia Spectrum Psychosis: Randomized, Parallel, Double- Blind, Placebo Controlled Trial
Brief Title: N-Acetyl-Cysteine (NAC) in Early Phase Schizophrenia Spectrum Psychosis
Acronym: NACPSY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Center de Neurosciences Psychiatrique, Lausanne, Switzerland (Unknown)
Responsible Party: Principal Investigator, Larry Seidman, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008P000460; 107865 (Other: FDA IND)
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenic Psychoses
Keywords: schizophrenia; schizoaffective; schizophreniform; early schizophrenia spectrum psychosis
MeSH Terms: conditions — Schizophrenia | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- n-acetyl-cysteine (Active Comparator): N-Acetyl cysteine effervescent tablets in water 2 in am and 1 in pm for 28 weeks
  Interventions: Drug: n-acetylcysteine
- Placebo (Placebo Comparator): matching effervescent tablets in water 2 in am and 1 in pm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: n-acetylcysteine — 900 mg effervescent PharmaNAC tablet in water or juice: two tablets in the AM, one tablet in PM
  Other Names: PharmaNAC
  Arms: n-acetyl-cysteine
Drug: Placebo — Placebo tablets are placed in water or juice in the AM and PM
  Arms: Placebo

SUMMARY:
The investigators seek to examine the effect of add-on N-Acetyl-Cysteine (NAC) in the early phase of schizophrenia spectrum illness in collaboration with researchers Kim Do, PhD, and Philippe Conus, MD in Switzerland. Modifications of brain structure are thought to occur during the pre-illness phase and around the transition to psychosis. Therefore, studying new treatments that could target changes occurring during this period is of critical importance.

Aims:

Does add-on NAC treatment in early psychosis influence:

* positive and negative symptoms
* extrapyramidal side-effects of other medication
* plasma concentration of glutathione
* Mismatch Negativity, a physiological marker

DETAILED DESCRIPTION:
The study proposes that a glutathione deficit leading to an abnormal response to oxidative stress is a vulnerability factor, combined with other brain specific factors, in brain functioning of some individuals with schizophrenia (Do et al., 2010). N-acetyl-cysteine is hypothesized to cross the blood-brain barrier and increase glutathione in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent
* DSM IV TR diagnosis of schizophrenia, schizophreniform, schizoaffective
* Psychiatric and medical stability
* Prescribing clinician's premission to participate, assurance of medical stability
* Having met threshold criteria for psychosis on CAARMS (Comprehensive Assessment of at Risk Mental States Scale) Psychosis subscale
* Up to 12 months of antipsychotic treatment

Exclusion Criteria:

* Severe medical comorbidities
* Previous cerebral trauma
* Substance induced psychosis or organic psychosis
* Mental retardation
* NAC allergy
* Pregnancy, females and males planning pregnancy
* Treatment with antioxidants
* Insufficient command of English

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Cousins, PhD, APRN, Study Director — Beth Israel Deaconess Medical Center; T. U. Wilson Woo, MD, PhD, Study Chair — Harvard Medical School (HMS and HSDM)
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts Mental Health Center, Boston, Massachusetts

REFERENCES:
- [Background] Do KQ, Conus P, Cuenod M. Redox dysregulation and oxidative stress in schizophrenia: nutrigenetics as a challenge in psychiatric disease prevention. World Rev Nutr Diet. 2010;101:131-153. doi: 10.1159/000314518. Epub 2010 Apr 30. No abstract available. PMID 20436260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at two sites, Lausanne University Hospital, Department of Psychiatry, Lausanne, Switzerland and at the Commonwealth Research Center of Beth Israel Deaconess Medical Center Boston, Massachusetts
Pre-assignment Details: 320 signed consent 133 declined to participate 124 excluded - 65 by Physician decision, 59 subject withdrew 63 met all inclusion and no exclusion criteria 31 to NAC and 30 to placebo
Groups:
- Placebo: matching effervescent tablets in water 2 in am and 1 in pm
  n-acetylcysteine: 900 mg effervescent PharmaNAC tablet in water or juice: two tablets in the AM, one tablet in PM
Period: Randomization
Arm/Group | N-acetyl-cysteine | Placebo
Started | 32 (1 never took study medication dropped by physician decision (White matter lesion on MRI)) | 31 (1 never took study medication due to subject withdrawal)
Completed | 31 | 30
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Double Blind (Visits 1-7)
Arm/Group | N-acetyl-cysteine | Placebo
Started | 31 (9 did not compete 7 study visits) | 30 (11 did not compete 7 study visits)
Completed More Than 1 Visit | 4 | 5
Stopped After First Visit | 3 | 2
Didn't Complete at Least 1 Visit | 2 | 4
Completed | 22 | 19
Not Completed | 9 | 11
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 8 | 11
Period: 1 Month Post Study Medication
Arm/Group | N-acetyl-cysteine | Placebo
Started | 22 | 19
1 Follow-up Visit (Visit 8) | 21 | 16
Completed | 21 | 16
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetyl-cysteine | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (6.1) | 24.7 (5.9) | 25.4 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 26 | 21 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 5 | 7 | 12
  White | 25 | 22 | 47
  Maghreb | 1 | 1 | 2
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 31 | 29 | 60
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 4 | 10
  Switzerland | 26 | 27 | 53
Positive and Negative Symptom Scale (PANSS) [Mean (Standard Deviation); unit: units on a scale] — Clinical Measure of Positive (7 items P1-P7) Negative Symptoms (7 items N1-N7) General Psychopathology Symptoms (G1-G16) total of 30 items
  Assessed in the previous week:
  RATING SCALE
  1: Absent 2: Minimal 3: Mild 4: Moderate 5: Moderate Severe 6: Severe 7: Extreme The higher the score the worse the symptoms. The lowest possible score is 30 and the highesr possible score is 210.
  units on a scale
    Positive PANSS Symptoms | 14.3 (5.4) | 15.0 (5.6) | 14.7 (16.4)
    Negative Symptoms | 15.6 (5.0) | 17.3 (6.3) | 16.4 (5.7)
Global Assessment of Functioning (GAF) [Mean (Standard Deviation); unit: units on a scale] — Clinical Measure of Global level of Symptoms (Sx) and Functioning from 1 (Worst) to 100 (Best) in groups of 10:
  100 - 91: Superior functioning 90 - 81: Absent or minimal Sx 80 - 71: If symptoms are present and expected 70 - 61:Some mild Sx 60 - 51: Moderate Sx 50 - 41: Serious Sx 40 - 31: Some impairment in reality testing or communication 30 - 21: Behavior is considerably influenced by delusions or hallucinations 20 - 11: Some danger of hurting self or others 10 - 1: Persistent danger of severely hurting self or others
  units on a scale | 54 (10.8) | 51.6 (12.8) | 52.8 (11.8)
Duration of Psychosis [Mean (Standard Deviation); unit: days] — Duration of time in days since onset of psychosis
  days | 848 (767) | 747 (693) | 796 (726)
Social and Occupational Functioning Assessment Scale (SOFAS) [Mean (Standard Deviation); unit: units on a scale] — Rating of Overall Social and Occupational Functioning on a scale of 1 (worst) to 100 (best) in groups of 10:
  100-91: Superior functioning 90-81: Good functioning 80-71: Slight impairment 70-61: Some difficulty 60-51: Moderate difficulty 50-41: Serious impairment 40-31: Major impairment 30-21: Inability to function in almost all areas 20-11: Unable to function independently 10-1: Unable to function without harming self or others
  units on a scale | 55.8 (11.0) | 53.5 (13.0) | 54.7 (12.0)
MATRICS Consensus Cognitive Battery (MCCB) excluding MISCEIT managing emotions test) [Mean (Standard Deviation); unit: Standardized T Scores] — The MCCB has 6 cognitive factors including: 1) processing speed (Trail Making Test, BACS: Symbol Coding, Category Fluency: Animal Naming), 2) sustained attention (Continuous Performance Test -Identical Pairs), 3) working memory (WMS-III Spatial Span and Letter-Number Span), 4) verbal learning (Hopkins Verbal Learning Test-Revised: Immediate Recall), 5) visual learning (Brief Visuospatial Memory test - Revised: Immediate Recall) and 6) problem solving (NAB Mazes). The T-score of 50 is an average score. Scores below 50 indicates cognitive processing lower than age matched healthy populations. Population: Numbers in each group analyzed based on those who completed baseline and post testing.
  Standardized T Scores
    Processing Speed: number analyzed (Participants) | 20 | 16 | 36
    Processing Speed | 37.72 (11.22) | 35.53 (16.31) | 36.75 (13.48)
    Sustained Attention: number analyzed (Participants) | 20 | 16 | 36
    Sustained Attention | 40.23 (11.71) | 32.67 (13.15) | 36.87 (12.35)
    Working Memory: number analyzed (Participants) | 20 | 16 | 36
    Working Memory | 47.56 (9.70) | 38.87 (15.09) | 43.70 (12.10)
    Verbal Learning: number analyzed (Participants) | 20 | 16 | 36
    Verbal Learning | 40.94 (10.09) | 40.93 (13.73) | 40.94 (11.71)
    Visual Learning: number analyzed (Participants) | 20 | 16 | 36
    Visual Learning | 41.06 (10.01) | 44.86 (14.42) | 42.75 (11.97)
    Problem Solving: number analyzed (Participants) | 20 | 16 | 36
    Problem Solving | 48.00 (11.69) | 39.93 (12.76) | 44.41 (12.17)
Antipsychotic Medication Chlorpromazine Equivalents [Mean (Standard Deviation); unit: milligrams] — Dose of current antipsychotic medication in chlorpromazine equivalents
  milligrams | 309 (252) | 309 (188) | 309 (220)
Blood Marker - Cysteine [Mean (Standard Deviation); unit: uM (micrometer)] — Cysteine is an amino acid, a building block for proteins and is used throughout the body and was measured in blood plasma.
  uM (micrometer) | 261.3 (37.6) | 254.0 (33.6) | 257.7 (35.7)
Blood Marker - GPxbc- Glutathione peroxidase [Mean (Standard Deviation); unit: umol/min/gHb] — GPxBC is a measurement of glutathiione peroxidase enzymatic activity in glutathione synthesis and the redox system in blood cells. Measured as umol/min/gHb from blood cells.
  umol/min/gHb | 21.24 (7.5) | 21.01 (6.93) | 21.13 (7.17)
Blood Marker - Glutathione [Mean (Standard Deviation); unit: mM (millimolar) in blood cells] — Glutathione is a tripeptide comprised of three amino acids (cysteine, glutamic acid, and glycine) and acts as an antioxidant, a free radical scavanger and a detoxifying agent. Glutathione is an important co-factor for the enzyme glutathione peroxidase used in the uptake of amino acids. The level of glutathione is measured in blood cells.
  mM (millimolar) in blood cells | 0.77 (0.21) | 0.84 (0.27) | 0.81 (0.24)
Brain Marker - Glutamine and myo-Inositol [Mean (Standard Deviation); unit: mM (millimolar)] — Brain levels of glutamine and myo-Inositol were measured using Magnetic ResonanceSpectroscopy (H-MRS), both are chemicals that work to protect the brain from high levels of excitatory chemicals such as glutamate. Population: MRS was completed on fewer participants.
  mM (millimolar)
    Glutamine: number analyzed (Participants) | 13 | 12 | 25
    Glutamine | 3.25 (0.51) | 2.93 (0.48) | 3.10 (0.50)
    Myo-Inositol: number analyzed (Participants) | 13 | 12 | 25
    Myo-Inositol | 6.25 (1.05) | 6.28 (0.62) | 6.26 (0.84)
Brain Marker - Glutathione and Glutamate [Mean (Standard Deviation); unit: mM (millimolar)] — Brain markers, glutathione and glutamate were measured using Magnetic Resonance Spectroscopy (H-MRS) in the medial prefrontal cortex. Glutathione is a tripeptide comprised of three amino acids (cysteine, glutamic acid, and glycine) and acts as an antioxidant, a free radical scavanger and a detoxifying agent. Glutathione is an important co-factor for the enzyme glutathione peroxidase used in the uptake of amino acids. Glutamate is an excitatory neurotransmitter in the brain. Population: Only 25 participants had the MRS.
  mM (millimolar)
    Glutathione: number analyzed (Participants) | 13 | 12 | 25
    Glutathione | 0.87 (0.23) | 1.12 (0.18) | 0.99 (0.21)
    Glutamate: number analyzed (Participants) | 13 | 12 | 25
    Glutamate | 10.12 (0.80) | 10.64 (1.23) | 10.37 (1.01)

OUTCOME MEASURES:

1. Primary Outcome: Change in Negative Symptoms of Schizophrenia as Measured on the PANSS
Description: Positive and Negative Symptom Scale was used to assess psychopathology. The sum of items N1 - N7 including N1) blunted affect, N2) emotional withdrawal, N3) poor rapport, N4) passive apathetic social withdrawal, N5) difficulty in abstract thinking, N6) lack of spontaneity and flow of conversation, and N7) sterotyped thinking were used to analyze negative symptoms of schizophrenia and were assessed for the previous week:
  RATING SCALE
  1: Absent 2: Minimal 3: Mild 4: Moderate 5: Moderate Severe 6: Severe 7: Extreme The higher the score the worse the symptoms. The lowest possible score is 7 and the highest possible score is 49 .
Time Frame: at 6 months
Population: Analysis was done with those who completed the 6 month treatment protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 22 | 19
units on a scale | 16.9 (4.9) | 17.2 (5.4)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.50, t-test, 2 sided

2. Secondary Outcome: Change in Positive Symptoms (PANSS)
Description: Positive and Negative Symptom Scale was used to assess psychopathology. The Positive symptom subscale of schizophrenia includes the sum of items P1 -P7 including P1) Delusions, P2) conceptual Disorganization, P3) Hallunicatory Behavior, P4) Excitement, P5) Grandiosity, P6) Suspiciousness and Persecution, and P7) Hostility and were assessed for the previous week:
  RATING SCALE
  1: Absent 2: Minimal 3: Mild 4: Moderate 5: Moderate Severe 6: Severe 7: Extreme The higher the score the worse the symptoms. The lowest possible score is 7 and the highest possible score is 49 .
Time Frame: at 6 months
Population: Analysis was done with participants who completed the 6 month treatment phase
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 22 | 19
units on a scale | 13.7 (7.8) | 12.5 (4.6)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.39, t-test, 2 sided

3. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: Measure Description: Clinical Measure of Global level of Symptoms (Sx) and Functioning from 1 (Worst) to 100 (Best) in groups of 10:
  100 - 91: Superior functioning 90 - 81: Absent or minimal Sx 80 - 71: If symptoms are present and expected 70 - 61:Some mild Sx 60 - 51: Moderate Sx 50 - 41: Serious Sx 40 - 31: Some impairment in reality testing or communication 30 - 21: Behavior is considerably influenced by delusions or hallucinations 20 - 11: Some danger of hurting self or others 10 - 1: Persistent danger of severely hurting self or others
Time Frame: at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 22 | 19
units on a scale | 52.2 (11.7) | 53.8 (11.6)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.52, t-test, 2 sided

4. Secondary Outcome: Social and Occupational Functioning Assessment Scale (SOFAS)
Description: Measure of social and occupational functioning using the Social and Occupational Functioning Assessment Scale Measure Description: Rating of Overall Social and Occupational Functioning on a scale of 1 (worst) to 100 (best) in groups of 10:
  100-91: Superior functioning 90-81: Good functioning 80-71: Slight impairment 70-61: Some difficulty 60-51: Moderate difficulty 50-41: Serious impairment 40-31: Major impairment 30-21: Inability to function in almost all areas 20-11: Unable to function independently 10-1: Unable to function without harming self or others
Time Frame: at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 22 | 19
units on a scale | 54.6 (11.3) | 54.8 (10.8)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.71, t-test, 2 sided

5. Secondary Outcome: Change in Cognition and Working Memory (MATRICS) Speed of Processing
Description: The MATRICS is neurocognitive battery designed to assess cognition. Processing speed is a composite score including the following tests: Trail Making Test, BACS: Symbol Coding, Category Fluency: Animal Naming. The score is a standardized T-Score which indicates the number of standard deviations above or below the mean, a T-Score of 50, in 10 point increments. A T-Score of 60 indicates 1 standard deviation above the mean and a T-Score of 40 indicates 1 standard deviation below the mean. A score below 50 indicated cognitive processing below that of an age and gender matched healthy control population. A score above 50 indicates cognitive processing above that of an age and gender matched healthy control population.
Time Frame: at 6 months
Population: Analysis of cognitive data is based on those who completed the cognitive testing at 6 months which required a separate clinic appointment and thus the overall number of participants is lower due to a loss of that data from failure to keep the cognitive testing appointment.
Measure: Mean (Standard Deviation); unit: T- Scores
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 20 | 16
T- Scores | 41.47 (11.45) | 35.85 (14.40)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Speed of Processing; Test type: Superiority; p = 0.022, t-test, 2 sided

6. Secondary Outcome: Change in Cognition and Working Memory (MATRICS) Working Memory
Description: The MATRICS is neurocognitive battery designed to assess cognition. Working Memory score is a composite score based on the following sub-test WMS-III Spatial Span and Letter-Number Span. The score is a standardized T-Score which indicates the number of standard deviations above or below the mean, a T-Score of 50, in 10 point increments. A T-Score of 60 indicates 1 standard deviation above the mean and a T-Score of 40 indicates 1 standard deviation below the mean. A score below 50 indicated cognitive processing below that of an age and gender matched healthy control population. A score above 50 indicates cognitive processing above that of an age and gender matched healthy control population.
Time Frame: at 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T- Scores
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 20 | 16
T- Scores | 47.47 (9.61) | 38.08 (17.70)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.270, t-test, 2 sided

7. Secondary Outcome: Change in Cognition and Working Memory (MATRICS) Attention and Vigilance
Description: The MATRICS is neurocognitive battery designed to assess cognition. Sustained attention and Vigilance is a composite score based on the Continuous Performance Test -Identical Pairs. The score is a standardized T-Score which indicates the number of standard deviations above or below the mean, a T-Score of 50, in 10 point increments. A T-Score of 60 indicates 1 standard deviation above the mean and a T-Score of 40 indicates 1 standard deviation below the mean. A score below 50 indicated cognitive processing below that of an age and gender matched healthy control population. A score above 50 indicates cognitive processing above that of an age and gender matched healthy control population.
Time Frame: at 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T- Scores
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 20 | 16
T- Scores | 40.92 (12.98) | 30.40 (13.91)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.153, t-test, 2 sided

8. Secondary Outcome: Change in Cognition and Working Memory (MATRICS) Verbal Learning
Description: The MATRICS is neurocognitive battery designed to assess cognition. Verbal Learning is a composite score based on the Hopkins Verbal Learning Test-Revised: Immediate Recall. The score is a standardized T-Score which indicates the number of standard deviations above or below the mean, a T-Score of 50, in 10 point increments. A T-Score of 60 indicates 1 standard deviation above the mean and a T-Score of 40 indicates 1 standard deviation below the mean. A score below 50 indicated cognitive processing below that of an age and gender matched healthy control population. A score above 50 indicates cognitive processing above that of an age and gender matched healthy control population.
Time Frame: at 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T- Scores
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 20 | 16
T- Scores | 42.18 (10.36) | 44.62 (12.34)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.876, t-test, 2 sided

9. Secondary Outcome: Change in Cognition and Working Memory (MATRICS) Visual Learning
Description: The MATRICS is neurocognitive battery designed to assess cognition. Visual Learning is a composite score based on the Brief Visuospatial Memory test - Revised: Immediate Recall. The score is a standardized T-Score which indicates the number of standard deviations above or below the mean, a T-Score of 50, in 10 point increments. A T-Score of 60 indicates 1 standard deviation above the mean and a T-Score of 40 indicates 1 standard deviation below the mean. A score below 50 indicated cognitive processing below that of an age and gender matched healthy control population. A score above 50 indicates cognitive processing above that of an age and gender matched healthy control population.
Time Frame: at 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T- Scores
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 20 | 16
T- Scores | 46.00 (9.28) | 47.75 (19.12)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.464, t-test, 2 sided

10. Secondary Outcome: Change in Cognition and Working Memory (MATRICS) Reasoning and Problem Solving
Description: The MATRICS is neurocognitive battery designed to assess cognition. Problem Solving is a composite score based on the NAB Mazes. The score is a standardized T-Score which indicates the number of standard deviations above or below the mean, a T-Score of 50, in 10 point increments. A T-Score of 60 indicates 1 standard deviation above the mean and a T-Score of 40 indicates 1 standard deviation below the mean. A score below 50 indicated cognitive processing below that of an age and gender matched healthy control population. A score above 50 indicates cognitive processing above that of an age and gender matched healthy control population.
Time Frame: at 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T- Scores
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 20 | 16
T- Scores | 51.13 (10.16) | 44.38 (12.80)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.741, t-test, 2 sided

11. Secondary Outcome: Change in Blood Level of Glutathione
Description: Glutathione is a tripeptide comprised of three amino acids (cysteine, glutamic acid, and glycine) and acts as an antioxidant, a free radical scavanger and a detoxifying agent. Glutathione is an important co-factor for the enzyme glutathione peroxidase used in the uptake of amino acids. The level of glutathione is measured in blood cells.
Time Frame: at 6 months
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 22 | 19
mM | 0.92 (0.42) | 0.82 (0.19)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.05, t-test, 2 sided

12. Secondary Outcome: Blood Plasma Level of Cysteine
Description: Cysteine is an amino acid, a building block for proteins and is used throughout the body and was measured in blood plasma.
Time Frame: at 6 months
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 22 | 19
uM | 229.6 (62.9) | 246.5 (42.4)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.33, t-test, 2 sided

13. Secondary Outcome: GPxbc Glutathione Peroxidase Activity in Blood Cells
Description: GPxBC is a measurement of glutathiione peroxidase enzymatic activity in glutathione synthesis and the redox system in blood cells. Measured as umol/min/gHb from blood cells.
Time Frame: at 6 months
Measure: Mean (Standard Deviation); unit: umol/min/gHb
Arm/Group | N-acetyl-cysteine | Placebo
Number analyzed (Participants) | 31 | 30
umol/min/gHb | 21.24 (7.5) | 21.01 (6.93)
Statistical Analysis 1: Comparison: N-acetyl-cysteine vs Placebo; Test type: Superiority; p = 0.90, t-test, 2 sided

14. Secondary Outcome: Glutamine Brain Level for NAC Group
Description: Glutamine is measured in the medial prefrontal cortex using Magnetic Resonance Spectroscopy (H-MRS) and is a chemical that works to protect the brain from high levels of excitatory chemicals such as glutamate.
Time Frame: at 6 months
Population: The number of subjects in the NAC and Placebo group is lower as not everyone in the study agreed to a MRS, in addition the MRS was only done at the Switzerland site.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | N-acetyl-cysteine
Number analyzed (Participants) | 13
mM | 3.16 (0.56)
Statistical Analysis 1: Comparison: N-acetyl-cysteine; Test type: Superiority; p = 0.6732, t-test, 1 sided

15. Secondary Outcome: Glutamine Brain Level for Placebo Group
Description: as for outcome 14
Time Frame: at 6 months
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mM
Groups:
- Placebo Group: Placebo comparison group for study matching effervescent tablets in water 2 in am and 1 in pm
  n-acetylcysteine: 900 mg effervescent PharmaNAC tablet in water or juice: two tablets in the AM, one tablet in PM
Arm/Group | Placebo Group
Number analyzed (Participants) | 12
mM | 2.90 (0.46)
Statistical Analysis 1: Comparison: Placebo Group; Test type: Superiority; p = 0.8786, t-test, 2 sided

16. Secondary Outcome: Glutamate Brain Level for NAC Group
Description: Brain marker, glutamate, was measured using Magnetic Resonance Spectroscopy (H-MRS) in the medial prefrontal cortex. Glutamate is an excitatory neurotransmitter in the brain.
Time Frame: at 6 months
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | N-acetyl-cysteine
Number analyzed (Participants) | 13
mM | 10.25 (1.20)
Statistical Analysis 1: Comparison: N-acetyl-cysteine; Test type: Superiority; p = 0.5622, t-test, 2 sided

17. Secondary Outcome: Glutamate Brain Level for Placebo Group
Description: as for outcome 14
Time Frame: at 6 months
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mM
Groups:
- Placebo Group: Placebo comparison group for study matching effervescent placebo tablets in water 2 in am and 1 in pm
Arm/Group | Placebo Group
Number analyzed (Participants) | 12
mM | 10.65 (1.26)
Statistical Analysis 1: Comparison: Placebo Group; Test type: Superiority; p = 0.9574, t-test, 2 sided

18. Secondary Outcome: Glutathione Brain Level for NAC Group
Description: measured by H-MRS in the medial prefrontal cortex Brain markers, glutathione was measured using Magnetic Resonance Spectroscopy (H-MRS) in the medial prefrontal cortex. Glutathione is a tripeptide comprised of three amino acids (cysteine, glutamic acid, and glycine) and acts as an antioxidant, a free radical scavanger and a detoxifying agent. Glutathione is an important co-factor for the enzyme glutathione peroxidase used in the uptake of amino acids.
Time Frame: at 6 months
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | N-acetyl-cysteine
Number analyzed (Participants) | 13
mM | 1.04 (0.27)
Statistical Analysis 1: Comparison: N-acetyl-cysteine; Test type: Superiority; p = 0.0043, t-test, 2 sided

19. Secondary Outcome: Glutathione Brain Level for Placebo Group
Description: as for outcome 18
Time Frame: at 6 months
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Placebo Group
Number analyzed (Participants) | 12
mM | 1.05 (0.20)
Statistical Analysis 1: Comparison: Placebo Group; Test type: Superiority; p = 0.3804, t-test, 2 sided

20. Secondary Outcome: Myo-Inositol Brain Level for the NAC Group
Description: Myo-Inositol is measured in the medial prefrontal cortex using Magnetic Resonance Spectroscopy (H-MRS)MRS and is a chemical that works to protect the brain from high levels of excitatory chemicals such as glutamate.
Time Frame: at 6 months
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | N-acetyl-cysteine
Number analyzed (Participants) | 13
mM | 6.27 (1.07)
Statistical Analysis 1: Comparison: N-acetyl-cysteine; Test type: Superiority; p = 0.9403, t-test, 2 sided

21. Secondary Outcome: Myo-Inositol Brain Level for Placebo Group
Description: as for outcome 20
Time Frame: at 6 months
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Placebo Group
Number analyzed (Participants) | 12
mM | 6.26 (1.05)
Statistical Analysis 1: Comparison: Placebo Group; Test type: Superiority; p = 0.9215, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline and 6 months
Description: Adverse Events were evaluated every month for 6 months and 1 month post treatment
Arm/Group | N-acetyl-cysteine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 26/31 | 29/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetyl-cysteine (N=31) | Placebo (N=30)
Tremor (Nervous system disorders) | 11 | 11
Rigidity (Nervous system disorders) | 7 | 13
Akathisia (Nervous system disorders) | 11 | 9
Dry Mouth (Nervous system disorders) | 16 | 15
Increased Salivation (Nervous system disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 10 | 11
Constipation (Gastrointestinal disorders) | 11 | 12
Hypotension (Cardiac disorders) | 7 | 8
Hypertension (Cardiac disorders) | 6 | 5
Emotional Indifference (Psychiatric disorders) | 17 | 21
Sedation (Nervous system disorders) | 18 | 21
Hair Loss (Skin and subcutaneous tissue disorders) | 4 | 4
Rash (Immune system disorders) | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No